CLINICAL TRIAL: NCT06574386
Title: Pregnancy in GUCH Patients: Maternal-Foetal-Neonatal Aspects at Mid Term
Brief Title: Pregnancy in GUCH Patients
Acronym: PURE-HEART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6487
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-08

CONDITIONS: Congenital Heart Disease; Pregnancy Related; Infant Development; IUGR; Fetal Growth Restriction
Keywords: GUCH; Pregnancy
MeSH Terms: conditions — Heart Defects, Congenital; Fetal Growth Retardation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Childhood neurodevelopment (Experimental): Newborns from mothers with congenital heart disease will be subjected to neurodevelopmental assessment
  Interventions: Diagnostic Test: Neurodevelopmental assessment

INTERVENTIONS:
Diagnostic Test: Neurodevelopmental assessment — Neurodevelopmental assessment

SUMMARY:
This study aims to investigate the impact of congenital heart diseases on maternal and foetal-neonatal health, the effect of pregnancy on maternal cardiac health, and the outcome of newborns/children born from Grown-Up Congenital Heart (GUCH) mothers with follow-up at one year, extendable to two.

The main question it aims to answer is:

-Does maternal congenital heart disease affects outcomes of newborn?

DETAILED DESCRIPTION:
After being informed about the study and potential risks all patients giving written informed consent will undergo:

* Cardiological and obstetric evaluation in the first trimester of pregnancy;
* Cardiological and obstetric revaluation in the second trimester of pregnancy;
* Cardiological and obstetric revaluation in the third trimester of pregnancy;
* Cardiac and general neonatal evaluation at birth;
* 2-year follow-up: maternal and neonatal cardiology evaluation, childhood neurodevelopment evaluation

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease in natural history or undergoing corrective and/or palliative cardiothoracic surgery.
* Chronological age > 18 years.
* Single pregnancy progressing normally at a gestational age of 14 weeks + 0.
* Correct pregnancy dating based on CRL as per ISUOG guidelines. (26)
* Normal results of non-invasive screening tests for foetal aneuploidies.
* Normal first-trimester ultrasound examination.
* Informed consent of the woman.

Exclusion Criteria:

* Maternal chromosomal abnormalities.
* Maternal syndromic conditions.
* Spontaneous abortion.
* Vanishing Twin.
* High risk for chromosomal abnormalities on screening tests performed in the 1st Trimester (Combined Test/NIPT) or Major foetal structural anomalies identified during first-trimester ultrasound evaluation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal outcomes in terms of weight and appropriate intrauterine development | Assessment in the first, second and third trimester of pregnancy
  Observation of neonatal outcome in terms of incidence of foetal growth restriction (FGR), defined as deviation from genetic potential with neonates classified as small for gestational age (SGA) or adequate for gestational age (AGA).

SECONDARY OUTCOMES:
Physical examination of the mother (BMI) | Assessment in the first, second and third trimester of pregnancy. Follow-up at 1 and 2 year from childbirth
  Physical examination will be evaluated by weight and height combination to report BMI in kg/m^2
Systolic and diastolic blood pressure of the mother during pregnancy | Assessment in the first, second and third trimester of pregnancy. Follow-up at 1 and 2 year from childbirth
  Systolic an diastolic blood pressure will be evaluated in mmHg
NYHA class progression during pregnancy (NYHA functional class) | Assessment in the first, second and third trimester of pregnancy. Follow-up at 1 and 2 year from childbirth
  NYHA class will be evalueted by medical examination during pregnancy
Cardiologic assessment of the mother (Electrocardiogram): | Assessment in the first, second and third trimester of pregnancy. Follow-up at 1 and 2 year from childbirth
  Cardiologic assesment will be evaluated by the use of Electrocardiogram (PR, QRS, QTc intervals and ST segment changes).
Cardiologic assesment of the mother (Echocardiography) | Assessment in the first, second and third trimester of pregnancy. Follow-up at 1 and 2 year from childbirth
  Cardiologic assesment will be evaluated by the use of echocardiography (wall motion assessment and residual congenital heart disease),
Cardiologic assesment of the mother (24-hour Holter ECG) | Assessment in the first, second and third trimester of pregnancy. Follow-up at 1 and 2 year from childbirth
  Cardiologic assesment will be evaluated by the use of 24-hour Holter ECG (ventricular and atrial arrhythmic burden)
Cardiologic assesment of the mother (24-hour Holter BP) | Assessment in the first, second and third trimester of pregnancy. Follow-up at 1 and 2 year from childbirth
  Cardiologic assesment will be evaluated by the use of 24-hour Holter BP (degree of arterial hypertension).
Assessment of foetal growth and weight (Subcutaneous Adipose Thickness SCAT) | Assessment in the first, second, third trimester of pregnancy, and at delivery. Follow-up at 1/2 years after delivery.
  Evaluated by abdominal adipose thickness index
Assessment of foetal oxygenation | Assessment in the first, second, third trimester of pregnancy, and at delivery. Follow-up at 1/2 years after delivery.
  Foetal oxygenation will be evaluated by rterial doppler of uterine arteries, umbilical arteries and middle cerebral artery and venous doppler of the umbilical vein and ductus venosus
Numbers of obstetric and maternal complications | Assessment in the first, second, third trimester of pregnancy, and at delivery. Follow-up at 1/2 years after delivery.
  Incidence of obstetric and maternal complications (maternal mortality, cardiac complications, hypertensive disorders, gestational diabetes, hepatosis, sepsis, placental abruption, thromboembolic events, postpartum haemorrhage, disseminated intravascular coagulation, need for further hospitalization; evaluation of mode of delivery)
Cardiological evaluation of the fetus | Assessment in the first, second, third trimester of pregnancy, and at delivery. Follow-up at 1/2 years after delivery.
  Cardiological evaluation of the fetus will be evaluated by foetal cardiotocography
Physical examination in newborns | Performed at birth, three months, and twelve months of age. Follow-up at 1/2 years after birth
  Physical examination will be evaluated by weight and height combination to report BMI in kg/m^2
Newborn's health and vital signs | At birth
  Evaluated by Apgar score calculation
Fetal metabolic condition | At birth
  Evaluated by umbilical artery blood gas analysis
Cardiologic assessment in newborns (Electrocardiogram) | Performed at birth, three months, and twelve months of age. Follow-up at 1/2 years after birth.
  Cardiologic assesment will be evaluated by the use of Electrocardiogram (PR, QRS, QTc intervals and ST segment changes).
Cardiologic assesment in newborns (Echocardiography) | Performed at birth, three months, and twelve months of age. Follow-up at 1/2 years after birth.
  Cardiologic assesment will be evaluated by the use of echocardiography (will be examined cardiac anatomical assessment; functional evaluation with left ventricular diastolic function and systolic function (EF and FS); right ventricular function; global function (MPI), PFO, PDA, pulmonary artery pressure, cardiac output, and input)
Neurological examination in newborns | Performed at birth, three months, and twelve months of age. Follow-up at 1/2 years after birth.
  Neurological evaluation will include cerebral ultrasound
Neurodevelopmental assessment in newborns (Hammersmith Infant Neurological Examination) | Performed at birth, three months, and twelve months of age. Follow-up at 1/2 years after birth.
  Neurological examination according to the Hammersmith Neonatal Neurological Examination
Physical growth in newborns (BMI) | Performed at birth, three months, and twelve months of age.
  Weight and height will be combined to report BMI in kg/m^2
Physical growth in newborns (head circumference in Cm) | Performed at birth, three months, and twelve months of age.
  It will be measured head circumference in centimeters
Respiratory function in newborns | Performed at birth, three months, and twelve months of age.
  Performed pulmonary function tests and nitrogen washout.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Massetti, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione universitaria policlinico Agostino Gemelli, Roma, Italy